CLINICAL TRIAL: NCT00511537
Title: Standard of Care Trial: Unrelated Stem Cell Transplantation for Adults With Hematopoietic Disorders
Brief Title: Unrelated Stem Cell Transplantation for Adults With Hematopoietic Disorders
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: UC-9907-CC99251
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: CML; ALL; AML; Myelodysplasia; Lymphoma; Myeloproliferative Disorders
Keywords: AML; ALL; CML; Lymphoma; Myelodysplasia; Unrelated stem cell transplantation; Hematopoietic disorders
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Lymphoma; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study performs HLA matched stem cell transplantation from unrelated donors in adults who require stem cell transplantation but do not have a matched related donor available. The incidence of graft-versus-host disease in unrelated stem cell transplantation is recorded. This study also monitors the activity and toxicity of total body irradiation and cyclosphosphamide followed by stem cell transplantation from matched unrelated donors.

DETAILED DESCRIPTION:
This protocol identifies a standard-of-care method for unrelated stem cell transplantation in adults. Performing this service in a consistent and documented fashion allows investigators to obtain informed consent from recipients. Data is tabulated locally for quality-control comparisons with nationally-reported standards. As a condition of maintaining transplant center status and to have acess to NMDP-registered donors, UCSF submits clinical and outcome data to the NMDP. As a result, UCSF is contributing to the resolution of remaining uncertainties regarding particular transplantation practices.

ELIGIBILITY:
Inclusion Criteria:

* Age >15 and <55
* Adequate renal function with serum creatinine <2.0 mg/dl
* Pulmonary diffusing capacity>50% of predicted
* Cardiac ejection fraction >40% as measured by radionuclide wall motion study or echocardiography
* Total bilirubin must be <2.5 mg/dl.
* Alkaline phosphatase and AST must be less than three times the upper limit of normal
* Negative serology for the human immunodeficiency virus
* Available HLA-matched donor
* Signed informed consent

Exclusion Criteria:

* No fully or single-antigen-mismatched sibling donor is available to donate stem cells
* No active liver disease.

Ages: 16 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Hematopoeietic Disorders
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 1999-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Martin, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States